CLINICAL TRIAL: NCT06160635
Title: D-SOLVE Cohorts (Cohort a and B)
Acronym: HDV750
Status: Recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: Karolinska University Hospital (Other); Karolinska Institutet (Other); Helmholtz Centre for Infection Research (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); National Institute of Infectious Diseases Matei Bals (Unknown)
Responsible Party: Sponsor
Other Study IDs: HDV750
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: HDV; HDV Infection; Chronic Liver Disease
Keywords: HDV; Hepatitis Delta; chronic liver disease; patient cohort; biomarker
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Biosamples: As part of the routine visit, structured biosampling for research purposes. Biosamples are collected as part of the clinical routine blood draw every 6 to 12 months. PBMC, plasma and samples for genetic studies are collected. Approximately 80 ml of additional blood is drawn.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Cohort A: Patients chronically infected with HDV. Patients with and without cirrhosis and with and without viremia will be included.
- Cohort B: Cohort B: Patients chronically infected with HDV and with available historical liver biopsies (5-20 years old biopsies) and clinical follow-up data or current patients willing to receive a core biopsy or fine-needle liver-cell aspirate (FNA). Patients with and without cirrhosis and with and without viremia will be included.

SUMMARY:
Hepatitis D is by far the most severe form of chronic viral hepatitis, frequently leading to liver failure, hepatocellular carcinoma and death. Hepatitis D is caused by coinfection Hepatitis D is caused by co-infection with hepatitis B virus (HBV) and hepatitis D virus (HDV).

This multicenter cohort should enable a comprehensive and unbiased biomarker screening of well-defined HDV-infected patients, followed by mechanistic studies to determine the functional role of distinct molecules. Patient surveillance strategies and antiviral treatment approaches could be personalized which should reduce clinical and social disease burden, improve quality of life and save direct and indirect costs caused by HDV infection.

DETAILED DESCRIPTION:
The D-SOLVE consortium ("Understanding the individual host response against Hepatitis D Virus to develop a personalized approach for the management of hepatitis D"), aims for an unbiased screening of a large multicenter cohort of well-defined HDV-infected patients to better understand individual factors determining the outcome of infection and to identify subjects benefitting from currently available treatments.

The D-SOLVE cohorts will be collected retrospectively as well as prospectively with clinical and virological data and biomaterial for the biomarker analysis. The aim of the cohorts is as following:

Cohort A: To define the demographic, clinical, virological, and immunological features of a large cross-sectional cohort of 750 untreated and treated HDV patients at 4 EU centers. To compare these features among patients with different origin, gender, disease severity and treatment. To collect biological material to generate translational studies, aimed to better understand pathogenesis, natural history and treatment response.

Cohort B: To identify histological and immunological features that are associated with fibrosis progression and clinical complications in patients with chronic HDV infection.

The D-SOLVE consortium has received funding from the Horizon 2020 EU Horizon Call "Personalised medicine and infectious diseases: understanding the individual host response to viruses (e.g. SARS-CoV-2)" of the European Union (grant agreement No 101057917). The consortium is coordinated by Hannover Medical School (MHH) and the Centre for Individualised Infection Medicine (CiiM). Other partners are:

* Helmholtz-Zentrum für Infektionsforschung (HZI), Germany
* Institut national de la santé et de la recherche médicale (INSERM)
* Karolinska Institutet (KI), Sweden
* Karolinska University Hospital / Region Stockholm (KUH), Sweden
* Policlinico of Milan (PFM), Italy
* National Institute for Infectious Diseases "Prof Dr Matei Balș" (INBIMB), Romania
* Helmholtz-Zentrum für Informationssicherheit (CISPA), Germany

The Cohorts and the biomarker screening are part of the EU-funded D-SOLVE Consortium.

ELIGIBILITY:
Inclusion Criteria:

* Anti-HDV positive
* ≥18 years old
* Sex: m/f/d
* Informed consent for prospective procedures

Exclusion Criteria:

* Anti-HDV negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients chronically infected with the hepatitis D virus (anti-HDV positive) can be included. For cohort B historical liver biopsies need to be available.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Biosample Screening | 3 years
  Identification of biomarkers that are associated with disease control, progression and treatment response by a multiomics approach that includes the investigation of: - the genome by the Illumina Infinium Global Screening array - the transcriptome by RNA-sequencing and single-cell RNA-sequencing (subset of samples) - the proteome by the Olink technology (high throughput proximity extension assay) - the metabolome by HPLC 1H-NMR (~2k metabolite features) - the methylome (Illumina 850k array) - immune phenotypes by high dimensional spectral flow cytometry - Spatial transcriptomics and multiplex imaging of HDV-patient liver biopsies

SECONDARY OUTCOMES:
Definition of the demographic, clinical and virological features of the cohort. | 3 years
  Identification of immunological determinants of liver disease progression, viral control and treatment response by - scRNA/ATAC sequencing of Ag-specific T cells, NK cells and MAIT cells (PBMC) - spatial multiomics with feature barcoding technology of liver core biopsies - Validation of findings by 29-color flow cytometry, hepatoma HDV infection system and respective mouse models
Identification of virological and immunological features and characteristics that relate to disease severity and treatment response. | 3 years
  Establishment of a computational model to predict immune responses and disease phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Markus Cornberg, Principal Investigator — Hannover Medical School
Locations (4):
- Hannover Medical School, Department of Gastroenterology, Hepatology, Infectious Disease and Endocrinology, Hanover, Germany
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico (University of Milan), Milan, Italy
- Institutul de Boli Infectioase "Prof. Dr. Matei Bals", Bucharest, Romania
- Karolinska University Hospital and Karolinska Institutet, Stockholm, Sweden